CLINICAL TRIAL: NCT07142720
Title: Clinical Study on Rapid Effects on Antioxidant Status, Immune Alertness, and Regenerative Activity
Brief Title: Rapid Effects on Antioxidant Status, Immune Alertness, and Regenerative Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Principal Investigator, Gitte Jensen, Ph.D., Principal Investogator, Natural Immune Systems Inc
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 176-005
Record Dates: First submitted 2025-08-13; First posted 2025-08-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Immune Surveillance; Stem Cell Surveillance

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blinded, cross-over study design.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will not be informed on which intervention they receive on any given day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Crossover group 1, randomized (Experimental): Crossover study: Participants consume a test product on each of the three clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume each of the 2 doses of the active test product versus placebo over 3 weeks. The order of interventions for this group is placebo, low dose, high dose.
  Interventions: Dietary Supplement: A low dose of seaweed extract; Dietary Supplement: A high dose of seaweed extract; Dietary Supplement: Placebo
- Crossover group 2, randomized (Experimental): Crossover study: Participants consume a test product on each of the three clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume each of the 2 doses of the active test product versus placebo over 3 weeks. The order of interventions for this group is low dose, high dose, placebo.
  Interventions: Dietary Supplement: A low dose of seaweed extract; Dietary Supplement: A high dose of seaweed extract; Dietary Supplement: Placebo
- Crossover group 3, randomized (Experimental): Crossover study: Participants consume a test product on each of the three clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume each of the 2 doses of the active test product versus placebo over 3 weeks. The order of interventions for this group is high dose, placebo, low dose.
  Interventions: Dietary Supplement: A low dose of seaweed extract; Dietary Supplement: A high dose of seaweed extract; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: A low dose of seaweed extract — A low dose of the seaweed extract is dissolved in plain rice milk to help camouflage the strong algae-taste.
Dietary Supplement: A high dose of seaweed extract — A high dose of the seaweed extract is dissolved in plain rice milk to help camouflage the strong algae-taste.
Dietary Supplement: Placebo — Plain rice milk.

SUMMARY:
This clinical study aims at documenting rapid effects after consuming single doses of test product, when compared to consuming a placebo.

A double-blind, placebo-controlled, cross-over study design will be used.

DETAILED DESCRIPTION:
For each participant, the clinic visits are scheduled at the same time of the day during the morning hours of 7-11 am to control for the effect of circadian fluctuations. One clinic visit involves consuming a placebo and serves as a control for the circadian variations in cytokine levels and immune surveillance for each participant. Since there is interference from exercise and stress with the release versus homing of lymphocytes, the study environment is managed so that any physical and mental stress is minimized during each visit. Upon arrival at a clinic visit, participants complete a questionnaire to help monitor exceptional circumstances that may influence the stress level of that person on that day. Predetermined criteria for re-scheduling a visit include sleep deprivation and acute anxiety. After completing the questionnaire, participants are instructed to remain calm and inactive for 3 hours, comfortably seated in a chair. After the first hour, the baseline blood sample is drawn. Immediately after the baseline sample is drawn, a test product is provided and consumed in the presence of clinic staff. Blood samples are drawn at 1 hour and 2 hours after consumption of the test product or placebo.

The blood is tested for antioxidant status, immune cell surveillance, and regenerating properties involving stem cell surveillance. The process of surveillance is the natural process of our immune and stem cells to move through our body and detect problems that need repair. In addition, blood samples are tested for changes to pro- and anti-inflammatory cytokines, antiviral peptides, and restorative growth factors.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults;
* Age 18-75 years (inclusive);
* Veins easy to see in one or both arms (to allow for the multiple blood draws);
* Willing to comply with a 24-hour wash-out period for vitamins and nutritional supplements;
* Willing to comply with study procedures, including:
* Maintaining a consistent diet and lifestyle routine throughout the study,
* Consistent habit of bland breakfasts on days of clinic visits,
* Abstaining from exercising and nutritional supplements on the morning of a study visit,
* Abstaining from use of coffee, tea, and soft drinks for at least one hour prior to a clinic visit;
* Abstaining from music, candy, gum, computer/cell phone use, during clinic visits.

Exclusion Criteria:

* Previous major gastrointestinal surgery (absorption of test product may be altered) (minor surgery not a problem, including previous removal of appendix and gall bladder);
* Taking anti-inflammatory medications on a daily basis;
* Currently experiencing intense stressful events/life changes;
* Currently in intensive athletic training (such as marathon runners);
* Currently taking antipsychotic medications such as clozapine, Risperdal, Abilify, Zyprexa or Seroquel;
* An unusual sleep routine (examples: working graveyard shift, irregular routine with frequent late nights, studying, partying);
* Unwilling to maintain a constant intake of supplements over the duration of the study;
* Anxiety about having blood drawn;
* Women of childbearing potential: Pregnant, nursing, or trying to become pregnant;
* Known food allergies related to ingredients in active test product or placebo.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Antioxidant uptake and protection | 1 and 2 hours
  Changes to antioxidant status of blood samples

SECONDARY OUTCOMES:
Immune cell numbers in blood | 1 and 2 hours
  Changes to immune cell trafficking and status of immune cell alertness, ie. the changes in immune cell populations and activation following consumption: Numbers of CD3- CD56+ NK cells in blood Numbers of CD3+ CD56+ NKT cells in blood Numbers of CD3+ CD56- T cells in blood Numbers of cells positive for CD25 Numbers of cells positive for CD69

OTHER OUTCOMES:
Stem Cell Numbers in Blood | 1 and 2 hours
  Changes to stem cell surveillance, i.e. the changes in stem cell populations following consumption of the study product: Numbers of CD45dimCD34+CD309+ pluripotential stem cells Numbers of Cd45dim CD34+CD309- progenitor stem cells Numbers of CD45-CD90+ lymphocytes in blood Numbers of CD31++ CD34- endothelial stem cells in blood
Communication through cytokines. | 1 and 2 hours
  Serum levels of cytokines, antiviral peptides, and restorative growth factors.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte S. Jensen, PhD, Principal Investigator — NIS Labs
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No